CLINICAL TRIAL: NCT03950505
Title: To Evaluate the Effect of Nesinaact on Non-alcoholic Steatohepatitis Through MRI and Liver Fibroscan in Patients With Type 2 Diabetes: A Prospective, Open-Label, Single-Arm, Single-Center Clinical Study
Brief Title: To Evaluate the Effect of Nesinaact on Non-alcoholic Steatohepatitis Through MRI and Liver Fibroscan in Patients With Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2018-0203
Record Dates: First submitted 2019-05-08; First posted 2019-05-15 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Non-alcoholic Steatohepatitis; Type2 Diabetes
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Pioglitazone; Therapeutics

STUDY DESIGN:
Intervention Model Description: This is a prospective, open-label, single-arm, single-center clinical Study. All participants will be treated with Nesinaact 25/15 (Alogliptin benzoate 25mg, pioglitazone hydrochloride 15mg) for 24 weeks.
Masking Description: No masking is applied, as this is an open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Nesinaact 25/15 (Alogliptin benzoate 25mg, pioglitazone hydrochloride 15mg) treatment for 24 weeks
  Interventions: Drug: Nesinaact 25/15 (Alogliptin benzoate 25mg, pioglitazone hydrochloride 15mg) treatment for 24 weeks

INTERVENTIONS:
Drug: Nesinaact 25/15 (Alogliptin benzoate 25mg, pioglitazone hydrochloride 15mg) treatment for 24 weeks — All participants will be treated with Nesinaact 25/15 (Alogliptin benzoate 25mg, pioglitazone hydrochloride 15mg) for 24 weeks. Patients who have not been prescribed any other anti-diabetic drugs at least for 12 weeks and whose HbA1c ranges from 6.5~8.5%, can be enrolled. If Patients has been prescribed metformin as monotherapy, they have to substitute metformin with nesinaact 25-15 for enrollment.

SUMMARY:
This study was designed to evaluate the effect of Nesinaact on non-alcoholic steatohepatitis through magnetic resonance imaging (MRI)-based proton density-fat fraction (MRI-PDFF) and liver fibroscan in patients with type 2 diabetes. This is a prospective, open-label, single-arm, single-center clinical Study. After 24 weeks of Nesinaact 25/15 (Alogliptin benzoate 25mg, pioglitazone hydrochloride 15mg) treatment, the improvement of parameters estimated by MRI and liver fibroscan will be estimated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ages >= 20 years
2. Patients diagnosed with non-alcoholic fatty liver disease (NAFLD).

   => Definition of NAFLD: CAP (Controlled attenuation parameter) >= 250 dB/m
3. Diabetic patients who meet one of the following glycemic conditions:

   * Patients with glycated hemoglobin (HbA1c) ranging 6.5~8.5 % while not taking an antidiabetic for more than 12 weeks irrespective of duration of diabetes.
   * Patients with HbA1c ranging 6.5~9.0 % in screening while using metformin monotherapy for more than 8 weeks without changing the dose irrespective of duration of diabetes.

Exclusion Criteria:

1. Patients who meet the criteria for alcoholic liver disease whose alcohol intake for the recent tow years if above 210 g per week in men and above 140 g per week in women)
2. Patients with chronic hepatitis B, C, or type 1 diabetes, or secondary diabetes
3. Patients with history of acute or chronic metabolic acidosis and ketoacidosis, including diabetic ketoacidosis accompanied or not accompanied by coma
4. Patients who were administered an oral hypoglycemic agent or insulin other than metformin within 8 weeks prior ro screening, or are likely to be administered it during the study duration among patients receiving monotherapy.
5. Patients who had hypersensitivity to biguanide or glitazone in the past.
6. Patients who received oral or parenteral corticosteroid treatment chronically (for more than 14 consecutive days) within 8 weeks prior to screening
7. Patients wih past history of lactic acidosis
8. Patients with a genetic disorder, such as galactose intolerance, Lapp lactase deficiency or glucose-galactose impaired absorption, etc.
9. Patients wih malnutrition, starvation, weakness, (Including patients with severe infection), pituitary insufficiency or adrenal insufficiency
10. Patients who have been receiving radiotherapy or chemotherapy due to bladder cancer and other malignant tumor, or it is less than 2 years since the patients received it.
11. Patients with past history of bladder cancer
12. A patient with history of drug abuse or alcoholism in 12 weeks
13. A patient who has hear failure (NYHA class 3~4) or uncontrolled arrhythmia within 6 months
14. A patient who has acute cardiovascular disease within 12 weeks (including unstable angina, myocardial infarction, transient ischemic attack, cerebrovascular disease, coronary artery bypass, or coronary intervention)
15. A person who falls under one of the followings:

1) A patient with serum creatinine level >= 1.5 mg/dL in men and 1.4 mg/dL in women or a patient wih moderate to severe renal impairment (creatinine clearance: < 50 ml/min) 2) An anemia patient with 10.5 g/dL of Hb level

* A pregnant or nursing woman
* A patient who does not consent to use a proper method of contraception during the study period only among women or men of childbearing age
* A patient who has taken investigational drug in other clinical study within 4 weeks following informed consent
* A person who may not participate in the study according to investigator's judgement
* A person who cannot read the informed consent form (e.g: an illiterate, a foreigner, etc.)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-05-29 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
A degree of liver steatosis | 24 weeks after starting Nesinaact 25/15 (Alogliptin benzoate 25mg, pioglitazone hydrochloride 15mg) treatment
  Magnetic resonance imaging (MRI)-based proton density-fat fraction (MRI-PDFF) will be evaluated to confirm the improvement in liver steatosis.
A degree of liver fibrosis | 24 weeks after starting Nesinaact 25/15 (Alogliptin benzoate 25mg, pioglitazone hydrochloride 15mg) treatment
  In liver fibroscan, liver stiffness (kPa) as a marker of fibrosis and CAP (dB/m) as a marker of steatosis will be estimated.

SECONDARY OUTCOMES:
Clinical glucometabolic parameters : HbA1c | 24 weeks after starting Nesinaact 25/15 (Alogliptin benzoate 25mg, pioglitazone hydrochloride 15mg) treatment
  HbA1c in %
Clinical glucometabolic parameters : Lipid parameters | 24 weeks after starting Nesinaact 25/15 (Alogliptin benzoate 25mg, pioglitazone hydrochloride 15mg) treatment
  Total cholesterol in mg/dL
Clinical glucometabolic parameters : Lipid parameters | 24 weeks after starting Nesinaact 25/15 (Alogliptin benzoate 25mg, pioglitazone hydrochloride 15mg) treatment
  Triglyceride in mg/dL
Clinical glucometabolic parameters : Lipid parameters | 24 weeks after starting Nesinaact 25/15 (Alogliptin benzoate 25mg, pioglitazone hydrochloride 15mg) treatment
  HDL-cholesterol in mg/dL
Clinical glucometabolic parameters : Lipid parameters | 24 weeks after starting Nesinaact 25/15 (Alogliptin benzoate 25mg, pioglitazone hydrochloride 15mg) treatment
  LDL-cholesterol in mg/dL
Clinical glucometabolic parameters : Liver enzymes | 24 weeks after starting Nesinaact 25/15 (Alogliptin benzoate 25mg, pioglitazone hydrochloride 15mg) treatment
  AST in IU/L
Clinical glucometabolic parameters : Liver enzymes | 24 weeks after starting Nesinaact 25/15 (Alogliptin benzoate 25mg, pioglitazone hydrochloride 15mg) treatment
  ALT in IU/L
Clinical glucometabolic parameters :Anthropometric parameters | 24 weeks after starting Nesinaact 25/15 (Alogliptin benzoate 25mg, pioglitazone hydrochloride 15mg) treatment
  Blood pressure in mmHg
Clinical glucometabolic parameters :Anthropometric parameters | 24 weeks after starting Nesinaact 25/15 (Alogliptin benzoate 25mg, pioglitazone hydrochloride 15mg) treatment
  Body weight in kilogram
Clinical glucometabolic parameters :Anthropometric parameters | 24 weeks after starting Nesinaact 25/15 (Alogliptin benzoate 25mg, pioglitazone hydrochloride 15mg) treatment
  Body mass idex in kg/m2

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Geriatrics, Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea